CLINICAL TRIAL: NCT03361384
Title: Alcohol and Implicit Process in Sexual Risk Behavior in MSM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Boston University (Other); University of South Dakota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-068; R01AA022301 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Drinking; Sex Behavior; Men
Keywords: men who have sex with men
MeSH Terms: conditions — Alcohol Drinking; Sexual Behavior; Multiple Endocrine Neoplasia Type 1; Homosexuality | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a beverage condition: alcohol, placebo, or control (water).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Alcohol condition (Experimental): The amount of alcohol received in the alcohol condition will be determined by an algorithm developed by Curtin (Curtin, 2000). Participants in the alcohol condition will receive a dose of alcohol (target BAC = .08%), administered in a chilled beverage of 80-proof vodka mixed with tonic water and lime juice in a 1:4 ratio.
  Interventions: Drug: Alcohol
- Placebo condition (Placebo Comparator): Placebo participants will receive tonic water and lime juice served to enhance alcohol cues in an amount comparable to the amount that they would have received if assigned to the alcohol condition.
  Interventions: Other: Placebo (non-alcoholic beverage)
- Control (water) (No Intervention): Participants in the water control condition will receive a glass of chilled water in volume of liquid comparable to the amount that they would have received if assigned to the alcohol or placebo condition.

INTERVENTIONS:
Drug: Alcohol
  Arms: Alcohol condition
Other: Placebo (non-alcoholic beverage)
  Arms: Placebo condition

SUMMARY:
The current study is the first empirical investigation that directly addresses the correspondence between responses regarding indicators of risky sexual behavior while under the influence of alcohol in the laboratory and the occurrence of sexually risky behavior while under the influence of alcohol in the natural environment, by use of Ecological Sampling Methodology (ESM). The study will allow us to compare and contrast implicit and explicit assessments of sexual risk in respect to future behavior in the natural environment. The data obtained will thus provide new information regarding the external validity of alcohol administration studies of sexual risk behavior and will provide information to optimize the selection of dependent measures. The current study also represents the first attempt to test a causal model linking alcohol intoxication and risky sexual behavior as a function of both automatic, reflexive, approach tendencies and effortful, deliberative, self-control (operationalized by executive working memory in this application). The ESM study will augment the findings of the experiment by providing a detailed assessment of contextual factors that affect sexual risk behavior as well as replicating and extending the findings of the experiment to sexual risk situations in the natural environment. Finally, to our knowledge there has been only one experimental study of alcohol and sexual risk in MSM (Maisto, Palfai, Vanable, Heath, & Woolf-King, 2012), which is remarkable given that MSM have been identified as the population at highest risk to contract the HIV in the U.S. since the virus was identified in the early 1980s. Thus the proposed research is only the second attempt to add to an understanding of the connections among alcohol, cognitive processes, and sexual risk behaviors in MSM.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 21-50
* Moderate or heavy drinkers based on classifications from the Quantity-Frequency-Variability Questionnaire (QFV; Cahalan, Cisin, & Crossley, 1969)
* Self-identify with the sexual orientation equivalent of a 3 or higher on the Kinsey Scale (Kinsey et al., 1948; Kinsey et al., 1953), a 7-point scale used to assess self-identified sexual orientation, with zero representing exclusive heterosexuality and 6 representing exclusive homosexuality.
* Participants must also have engaged in sex with other men at least once/month for the past 3 months.

Exclusion Criteria:

* a) under the age of 21 or b) do not have a government issued ID or c) are not able to provide medical records or other official documents with a birthdate (e.g., birth certificate), accompanied by a photo ID
* Scores ≥ 5 on the Brief Michigan Alcoholism Screening Test (Brief MAST; Pokorny, Miller, & Kaplan, 1972)
* Any ASSIST substance involvement score of ≥ 27 (National Institute on Drug Abuse; http://www.drugabuse.gov/sites/default/files/pdf/nmassist.pdf)
* Score ≥ 15 on the Patient Health Questionnaire-8 (PHQ-8; Kroenke et al., 2009)
* 4 subscales of the Brief Symptom Inventory (BSI; Derogatis & Melisaratos, 1979), Somatization, Obsession-compulsion, Paranoid ideation, and Psychoticism will be administered; Individuals experiencing severe psychological health symptoms (score > 2 on any item) will be further questioned by a research assistant in order to determine if there is psychiatric distress or problems present
* Report current medications or current medical problems (e.g., liver disorders, heart disease, HIV+ serostatus) that contraindicate alcohol use using the Medical Condition Questionnaire; Participants who confirm that they are using (i.e., have used in the past week) any prescribed drugs for which alcohol use is contraindicated (http://www.nlm.nih.gov/medlineplus/druginfo/drug_Aa.html) will be excluded. Participants also currently regularly taking (i.e., past 24 hours) any herbals and vitamins, including sleep aids (chamomile) and herbal preparations for anxiety and depression (Kava Kava or St. John's Wort) that contraindicate alcohol use will be excluded
* Persons with cognitive and or psychomotor deficits will be excluded from the experiment (based on RA and PI determination)
* Endorse currently being in a committed, exclusive monogamous relationship
* Report treatment for emotional or substance use disorders (defined by current treatment or treatment in the past 3 months) or recent history of significant alcohol problems as indicated by inpatient/outpatient alcohol treatment or alcohol self-help group attendance (e.g., AA) within the past 3 years.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 260 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Risk exposure | Post beverage administration (completed 30-45 minutes following beverage consumption)
  Behavioral skills and risk exposure will be measured with two interactive videos developed for the Maisto et al. (2012) experiment. For the risk exposure component, each video begins by setting a scene in which "Jim" (the protagonist) and "Dave" (the character with whom the participant will be asked to identify) meet up with each other. The participant will be asked to make a series (5 choice points) of binary choices (yes/no) about engaging in various increasingly high-risk sexual activities with Jim. Participants will receive 1 point for each time they answer "yes" and thus make a progressively risky choice. The risk exposure portion of the video will terminate with the first "no" response to the choice points. Subsequently, the participant will go to the fifth choice point to begin the behavioral skills component of the video. The risk exposure score will represent the mean score from the two interactive videos. Higher scores represent higher risk exposure scores.
Behavioral skills | Post beverage administration (completed 30-45 minutes following beverage consumption)
  The behavioral skills portion of the video will require participants to negotiate sexual situations using verbal communication skills in an interactive role-play. Participants will be asked to respond first to Jim's comment that he desires to have unprotected anal sex and that there is no cause for concern because he is safe ("prompt 1") and = a second, more insistent comment that was a reminder to the participant that UAI would not be risky and would be pleasurable and that the participants could trust Jim ("prompt 2"). Participants' responses to each of the prompts will be scored on a 0-2 scale (higher score = better communication skills). The behavioral skills score will represent the mean score from the two interactive videos.
Intentions to engage in unprotected sex | Post beverage administration (completed 30-45 minutes following beverage consumption)
  Intention to engage in unprotected sex after viewing each of two sexual video vignettes (Maisto et al., 2012) will be rated on a 7-point rating scale (Bishop & Maisto, 2011). The intentions to engage in unprotected sex score will represent the mean score from the two interactive videos. Higher scores represent greater intentions to engage in unprotected sex.

CONTACTS AND LOCATIONS:
Overall Officials: Steve A Maisto, PhD, Principal Investigator — Syracuse University; Jeffrey Simons, PhD, Principal Investigator — University of South Dakota; Tibor P.A. Palfai, PhD, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - Boston University, Boston, Massachusetts
  - Syracuse University, Syracuse, New York
  - University of South Dakota, Vermillion, South Dakota

IPD SHARING:
Plan to Share IPD: Undecided